CLINICAL TRIAL: NCT06451120
Title: Study of Platelet Rich Plasma (PRP) Injections With Symptomatic Knee Osteoarthritis for Biomarker Exploration in Young and Old Human Subjects
Brief Title: Platelet Rich Plasma Injections In Young And Old Human Subjects
Acronym: PRP-KOBE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 22-38279
Record Dates: First submitted 2024-05-30; First posted 2024-06-11 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Osteoarthritis; Articular Cartilage; Musculoskeletal Disorders
Keywords: Platelet-rich plasma (PRP)
MeSH Terms: conditions — Osteoarthritis; Musculoskeletal Diseases | interventions — Injections; Prolactin-Releasing Hormone

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-blind, placebo-controlled trial with a secondary crossover phase at the end of the initial trial to ensure all subjects receive one PRP injection. The randomization will be stratified by two age groups (ages 18-45 yrs. and 46-70 yrs).
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Platelet-rich plasma (PRP) (Experimental): A vacutainer vial containing 50 mL of peripheral blood will be processed immediately to create PRP using a previously optimized two-step centrifugation protocol viii. First, the whole blood will be centrifuged at 500 x g for 8 minutes at 4°C. The plasma will be collected above the buffy coat using a sterile pipette, placed into a separate sterile tube, and centrifuged a second time at 700 x g for 17 minutes at 12° C. The top 70% will be collected as the PPP and the bottom 30% will be resuspended as the PRP. PPP will be aliquoted into cryovials for storage at -80 °C. Approximately 6 mL of PRP will be produced from each 50 mL vial of whole blood. Five mL will be allocated for administration to patients and the remaining one mL will be aliquoted into cryovials for storage at -80 °C. The syringe containing PRP will be covered with Aluminum foil, such that the investigator cannot tell what fluid is to be injected.
  Interventions: Drug: Platelet-Rich Plasma (PRP) Injections; Device: Centrifuge
- Control saline injection (wait-list control) (Placebo Comparator): A placebo injection of 6 mL of 0.9% saline will be prepared by the unblinded research assistant in an adjacent room. The syringed will be prepared in a 10 mL syringe and covered with Aluminum foil, such that the investigator performing the injection cannot tell if there is PRP or saline to be injected.
  Interventions: Drug: Platelet-Rich Plasma (PRP) Injections; Drug: Control saline injection

INTERVENTIONS:
Drug: Platelet-Rich Plasma (PRP) Injections — Bloods will be drawn prior to the PRP injection, and repeated at 2 weeks, 12 weeks, possibly 14 weeks for crossover patients follow up visits. Under aseptic technique with a surgical drape/curtain in place to block the study subject's view of the knee. Syringes will be covered with aluminum foil and subjects will have a cover over their eyes, so that neither subjects nor the clinical investigator will know if the injection delivered is PRP injection or a normal saline injection
  Other Names: platelet-rich growth factors (GFs), platelet-rich fibrin (PRF) and platelet concentrates (PCs)
Device: Centrifuge — The Eppendorf Centrifuge is used to make the PRP. In our opinion, the centrifuge is a nonsignificant risk device. The centrifuge, sterile vials for blood collection and PRP injection syringes do not present a potential risk for serious health, safety or welfare of a subject. It is not needed to support or sustain human life. It is not of substantial importance in diagnosis, curing, mitigating or treating disease for the health, safety and welfare of the patients. There are no potential for serious risk to the health, safety or welfare of a subject.
  Other Names: Microcentrifuge tubes, Eppendorf tubes
  Arms: Platelet-rich plasma (PRP)
Drug: Control saline injection — A placebo injection of 6 mL of 0.9% saline will be prepared by the unblinded research assistant in an adjacent room. The syringed will be prepared in a 10 mL syringe and covered with Aluminum foil, such that the investigator performing the injection cannot tell if there is PRP or saline to be injected.
  Arms: Control saline injection (wait-list control)

SUMMARY:
This is a randomized, double-blind, placebo-controlled phase 2 study with a secondary crossover phase at the end of the initial trial to ensure all subjects receive one PRP injection. The goal is to identify what proteins change in the blood following repeated intraarticular knee PRP injections in patients with knee osteoarthritis. The objective is to determine the protein changes resulting from a single autologous PRP injection (5 mL) in comparison to a normal saline control.

About 60 subjects will take part in this study by two age groups at UCSF into the following arms: Arm A: PRP injection; Arm B: normal saline injection control. The study aims to demonstrate what benefits PRP has on knee osteoarthritis and methods to best achieve biologic effects. Subjects with a diagnosis of knee osteoarthritis ages 18-45 and 46-70 years old presenting to a University Based sports medicine clinic will be screened for potential eligibility. Subjects who meet all qualifying requirements will be recruited from UCSF's orthopedic and primary care clinics.

Subjects will be on study for up to 26 weeks Screening: up to 14 days Treatment: injection of PRP or normal saline; subjects can cross over at week 12 to a PRP if originally in the control injection group Follow-up: 2 weeks post-baseline injection, 12 weeks postbaseline, (14 weeks if crossover patient), 26 weeks.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled trial with a secondary crossover phase at the end of the initial trial to ensure all subjects receive one PRP injection. The randomization will be stratified by two age groups (ages 18-45 yrs. and 46-70 yrs).Screening and medical chart data will be reviewed to determine subject eligibility.

Platelet rich plasma (PRP) falls under transfusion medicine which has been FDA approved. Seeking to identify biological pathways by which PRP acts in a degenerative condition like knee osteoarthritis. The study compares the immediate and delayed variations in blood and synovial fluid biomarkers following PRP knee intraarticular injections in younger and older patients with knee osteoarthritis. The differences in blood biomarkers between ages of Knee osteoarthritis (KOA) patients are being investigated in this study. Intra-individual variations in some blood proteins will deviate (e.g., be larger or lower) from a normal saline control between week two and week twelve following the 5 mL PRP injection.

The unblinded research evaluation will evaluate the first batch of the first 20 blood and synovial fluid samples to ensure that the tests provide the desired results and data outcomes.

The visits consist of the Baseline visits (Week 0), the Week 2 visit, and the Week 12 visit and for half of the participants an optional 14 Week visit. These are in person visits. There are three remote visits at Week 26, Week 52 and Week 104.

Participation is estimated to take 2-2.5 hours for each visit over 6 months. The time it takes for each participant to attend an on-site visit is approximately 2-2.5 hours in total each time. The knee injection takes approximately 45 minutes for blood or knee fluid donation and preparation of the PRP. This injection occurs 1-2 times, depending on randomization arm). Subjects will complete surveys at the 3-4 timepoints, estimated to take 30 minutes per timepoint (or total); perform functional testing which is walking 40 meters back and forth quickly, sitting and standing for 30 seconds, and climbing stairs for 3 minutes and have the activity monitor put on (15 minutes). Subject will complete study questionnaires at the beginning of each visit (30 minutes). In addition, participants are asked to engage in physical therapy ideally once a week for 10 weeks although this will be documented as it is standardized but not required for the study.

If subjects are assigned to the Placebo Arm (Arm B), subjects will be informed that of receiving the placebo (normal saline injection) rather than the PRP injection. Subject will be offered the option of crossing over to receive a PRP injection. If a subject agrees to have a PRP injection, researchers will collect research blood (about 60cc or 4 tablespoons) and fluid from the knee joint space. If the subject decides to receive the PRP injection, the researchers will collect research blood (approximately 20ml or 1.5 tablespoons) and fluid from the knee joint space (45 minutes). The subject will fill out a questionnaire (30 minutes) and perform tasks to test their function (45 minutes). At the baseline appointment, subjects will receive an activity monitor to use for one week. The activity monitor should be returned on the week 14 visit.

Week 14 on site visit - If subjects are given a PRP injection at 12 weeks, subjects will have a two-week follow-up visit. The researchers will collect research blood (about 20ml or 2 tablespoons) and fluid from the knee joint space. Subjects will complete a questionnaire, and tasks testing the subject's function. Subjects will go home with an activity monitor that subjects will be asked to wear for 1 week. The activity monitor should be returned. Subjects will be asked to keep a diary to record symptoms and pain medication intake following injections. The participants will be interviewed and have their diaries reviewed on follow up visits.

ELIGIBILITY:
Inclusion Criteria

1. Grade 1-3 KL score will be recruited;
2. Symptoms of knee osteoarthritis for at least 3 months before presentation in one knee;
3. Have symptomatic complaints from osteoarthritis pain in no other joint affecting the hips, ankles or unaffected knee;
4. Will be able to attend and perform physical therapy.
5. English-speaking

Exclusion Criteria

1. Patients will be excluded if:

1. Received injection therapy for knee osteoarthritis in the past 6 months
2. Have signs of concomitant osteoarthritis of 1 or more other major joints of the lower extremities that impair their daily activity level
3. History of septic arthritis
4. Have underwent a previous knee surgery specifically for osteoarthritis or osteochondral defects less than 1 year before randomization (i.e. autograft or allograft surgery
5. High tibial osteotomy, partial knee replacement, patellar resurfacing), total knee replacement or existing surgical hardware in the knee
6. Patient with platelet disorders, bleeding disorder
7. Patient with rheumatologic disease, automimmune disorder, immunocompromised status, active history of cancer
8. Patient taking Chemotherapy, need for regular prednisone or antiinflammatory used
9. Pregnant, breastfeeding, or unwilling to practice birth control during participation in the study.
10. Uncontrolled illness, physical disability, or other contraindication to aerobic exercise training including, but not limited to:

i. Acute myocardial Infarction (within 5 days of any planned study procedure); ii. Unstable angina; iii. Uncontrolled arrhythmia causing symptoms or hemodynamic compromise; iv. Recurrent syncope; v. Active endocarditis; vi. Acute myocarditis or pericarditis; vii. Symptomatic severe aortic stenosis; viii. Uncontrolled heart failure; ix. Acute (within 3 months) pulmonary embolus or pulmonary infarction; x. Thrombosis of lower extremities; xi. Suspected dissecting aneurysm; xii. Uncontrolled asthma; xiii. Pulmonary edema; xiv. Room air desaturation at rest ≤85%; xv. Respiratory failure; xvi. Acute non-cardiopulmonary disorders that may affect exercise performance or be aggravated by exercise (ie infection, renal failure, thyrotoxicosis); and xvii. Mental impairment leading to inability to cooperate.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-12-18 (Estimated); Study Completion 2025-12-18 (Estimated)

PRIMARY OUTCOMES:
Identify Protein Changes in Platelet Rich Plasma (PRP) | 2 weeks
  The protein changes from a single autologous PRP injection (5 mL) vs normal saline control, using proteomic analysis of' venous blood samples. For proteomic analysis of Platelet poor plasma (PPP) and PRP, the samples will undergo quantitative mass spectrometry, with higher numbers indicating more proteins and lower numbers meaning less proteins.

SECONDARY OUTCOMES:
To determine the Intra-individual change in specific proteins in the peripheral blood | 12 weeks
  Changes in specific proteins in the blood will be different (e.g., higher or lower) after the 5 mL PRP injection compared to a normal saline control using proteomic analysis. PPP and PRP samples will undergo quantitative mass spectrometry, with higher numbers indicating more proteins and lower numbers meaning less proteins.

OTHER OUTCOMES:
To determine the Protein Changes in the synovial vluid | 2 weeks and 12 weeks
  Using proteomic analysis of the synovial fluid at the knee, compare the protein alterations caused by an autologous PRP dose (5 mL) to the normal saline control. For proteomic analysis of synovial fluid, the samples will undergo quantitative mass spectrometry, with higher numbers indicating more proteins and lower numbers meaning less proteins.
Examine Differences by Age | 2 weeks and 12 weeks
  Protein alterations in blood and synovial fluid following knee injections. For each arm, investigator will compare groups of young people (18-45 years old) and older people (46-70 years old) independently.
Change in Visual Analog Pain Scores | 2 weeks, 12 weeks and 26 weeks
  Pain will be measured using the Visual Analog Pain Scores, the score ranges from 0-10, zero indicating no pain and 10 being the worst pain ever.
Changes in Knee Injury and Osteoarthritis Outcome Scores (KOOS scores) | 2 weeks, 12 weeks and 26 weeks
  Knee Injury and Osteoarthritis Outcome Scores (KOOS scores), the score ranges from 0-100, with 0 representing extreme knee problems and 100 representing no knee problems.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Luke, MD, MPH, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Van Blarigan EL, Kenfield SA, Olshen A, Panchal N, Encabo K, Tenggara I, Graff RE, Bang AS, Shinohara K, Cooperberg MR, Carroll PR, Jones LW, Winters-Stone K, Luke A, Chan JM. Effect of a Home-based Walking Intervention on Cardiopulmonary Fitness and Quality of Life Among Men with Prostate Cancer on Active Surveillance: The Active Surveillance Exercise Randomized Controlled Trial. Eur Urol Oncol. 2024 Jun;7(3):519-526. doi: 10.1016/j.euo.2023.10.012. Epub 2023 Oct 29. PMID 37907387
- [Background] Schroer AB, Ventura PB, Sucharov J, Misra R, Chui MKK, Bieri G, Horowitz AM, Smith LK, Encabo K, Tenggara I, Couthouis J, Gross JD, Chan JM, Luke A, Villeda SA. Platelet factors attenuate inflammation and rescue cognition in ageing. Nature. 2023 Aug;620(7976):1071-1079. doi: 10.1038/s41586-023-06436-3. Epub 2023 Aug 16. PMID 37587343
- [Background] Van Blarigan EL, Chan JM, Sanchez A, Zhang L, Winters-Stone K, Liu V, Macaire G, Panchal N, Graff RE, Tenggara I, Luke A, Simko JP, Cooperberg MR, Carroll PR, Kenfield SA. Protocol for a 4-arm randomized controlled trial testing remotely delivered exercise-only, diet-only, and exercise + diet interventions among men with prostate cancer treated with radical prostatectomy (Prostate 8-II). Contemp Clin Trials. 2023 Feb;125:107079. doi: 10.1016/j.cct.2023.107079. Epub 2023 Jan 5. PMID 36621597
- [Background] Langlais CS, Chen YH, Van Blarigan EL, Chan JM, Ryan CJ, Zhang L, Borno HT, Newton RU, Luke A, Bang AS, Panchal N, Tenggara I, Schultz B, Lavaki E, Pinto N, Aggarwal R, Friedlander T, Koshkin VS, Harzstark AL, Small EJ, Kenfield SA. Quality of life for men with metastatic castrate-resistant prostate cancer participating in an aerobic and resistance exercise pilot intervention. Urol Oncol. 2023 Mar;41(3):146.e1-146.e11. doi: 10.1016/j.urolonc.2022.11.016. Epub 2022 Dec 15. PMID 36528473
- [Background] Kenfield SA, Van Blarigan EL, Panchal N, Bang A, Zhang L, Graff RE, Chen YH, Ryan CJ, Luke A, Newton RU, Tenggara I, Schultz B, Wang E, Lavaki E, Zuniga K, Pinto N, Borno H, Aggarwal R, Friedlander T, Koshkin VS, Harzstark A, Small E, Chan JM. Feasibility, safety, and acceptability of a remotely monitored exercise pilot CHAMP: A Clinical trial of High-intensity Aerobic and resistance exercise for Metastatic castrate-resistant Prostate cancer. Cancer Med. 2021 Nov;10(22):8058-8070. doi: 10.1002/cam4.4324. Epub 2021 Oct 12. PMID 34636156
- [Background] Tangtiphaiboontana J, Figoni AM, Luke A, Zhang AL, Feeley BT, Ma CB. The effects of nonsteroidal anti-inflammatory medications after rotator cuff surgery: a randomized, double-blind, placebo-controlled trial. J Shoulder Elbow Surg. 2021 Sep;30(9):1990-1997. doi: 10.1016/j.jse.2021.05.018. Epub 2021 Jun 24. PMID 34174448
- [Background] Lazaro RM, Souza RB, Luke AC. Patellar mobility and lower limb kinematics during functional activities in individuals with and without patellar tendinopathy. Knee. 2021 Jun;30:241-248. doi: 10.1016/j.knee.2021.04.002. Epub 2021 May 3. PMID 33957465
- [Background] Krabak BJ, Roberts WO, Tenforde AS, Ackerman KE, Adami PE, Baggish AL, Barrack M, Cianca J, Davis I, D'Hemecourt P, Fredericson M, Goldman JT, Harrast MA, Heiderscheit BC, Hollander K, Kraus E, Luke A, Miller E, Moyer M, Rauh MJ, Toresdahl BG, Wasfy MM. Youth running consensus statement: minimising risk of injury and illness in youth runners. Br J Sports Med. 2021 Mar;55(6):305-318. doi: 10.1136/bjsports-2020-102518. Epub 2020 Oct 29. PMID 33122252
- [Background] Lau BC, Motamedi D, Luke A. Use of Pocket-Sized Ultrasound Device in the Diagnosis of Shoulder Pathology. Clin J Sport Med. 2020 Jan;30(1):20-24. doi: 10.1097/JSM.0000000000000577. PMID 31855908
- [Background] Mah CD, Sparks AJ, Samaan MA, Souza RB, Luke A. Sleep restriction impairs maximal jump performance and joint coordination in elite athletes. J Sports Sci. 2019 Sep;37(17):1981-1988. doi: 10.1080/02640414.2019.1612504. Epub 2019 May 24. PMID 31122131